CLINICAL TRIAL: NCT02793791
Title: Prophylactic Minimally-invasive Local Ablation Therapies for the Hepatic Dysplastic Nodules in Patients With Positive Hepatitis B Surface Antigen (HBsAg).
Brief Title: Prophylactic Treatment of Hepatic Dysplastic Nodules in HBsAg Positive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Lei ZHAO, Doctor; Director, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDCHI-HDN
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Dysplastic Nodule of Liver; Chronic Hepatitis B
Keywords: high grade dysplastic nodule (HGDN); low grade dysplastic nodule (LGDN)
MeSH Terms: conditions — Hepatitis B, Chronic

ARMS (2):
- Ablation (Experimental)
  Interventions: Procedure: minimally invasive ablation therapies
- Observation (No Intervention)

INTERVENTIONS:
Procedure: minimally invasive ablation therapies — Including RFA (radiofrequency ablation);MWA (microwave ablation); PEI (percutaneous ethanol injection),etc.
  Arms: Ablation

SUMMARY:
The aim of this study is to determine that for hepatic dysplastic nodules in patients with chronic hepatitis B, instead of enhanced follow-up, whether early minimally-invasive ablation therapy can reduce the incidence of hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatic dysplastic nodules (DNs) include high grade dysplastic nodules (HGDNs) and low grade dysplastic nodule (LGDNs), their incidences are high in patients with liver cirrhosis. Once diagnosed, all latest versions of the major guidelines recommend enhanced follow-up, and no treatment would be provided until the diagnosis of hepatocellular carcinoma (HCC) is established during the follow-up.

While on the other hand, mounting evidence shows that DNs have relatively high transition rate to progress to HCC. In 154 patients with chronic hepatitis and cirrhosis, Kobayashi et al. reported the annual transition rate of 20% for patients with HGDN and 10% for patients with LGDN. The 5-year cumulative transition rate from HGDN and LGDN was 80.8% and 30.2%, respectively. Even regenerative nodules (RNs) without dysplasia evolved into HCC in 12.4%.More recently, Sato et al. studied 68 large regenerative nodules (LRNs) and 20 DNs from 1,500 consecutive nodular lesions; the 50-month transition rate was 13.6% in LRNs and 40% in DNs. Earlier studies support these findings.

Adenomatous polyps are accepted precursors to colorectal cancer (CRC) and removed to prevent cancer. Compared to the above transition rates, A recent cohort study estimated that the average annual transition rate from advanced adenoma to CRC in men was 3.1%,so the 5-year-transition rate was around 15%. Since the transition rate of hepatic DNs is much higher than the colorectal adenomatous polyps, is "enhanced follow-up" really the best choice of the treatment?

So in this proposed clinical trial, we hypothesize that for hepatic DNs discovered in patients with chronic hepatitis B, early minimally-invasive ablation treatment will decrease the incidence of HCC.

Recruited patients will be divided in to two groups randomly, in the "Observation group", patients will be followed-up and receive no therapy; while in the "Ablation group", the DNs will be ablated by minimally-invasive ablation therapies, including RFA, PEI, MWA, etc. All patients will be followed-up according to the AASLD guideline. Then the incidence of HCC of the two arms will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HBV
* Diagnosis of hepatic dysplastic nodule(s) be confirmed by biopsy.

Exclusion Criteria:

* concurrent HCV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatocellular carcinoma during the follow-up | Up to 70 months
  The diagnosis of hepatocellular carcinoma during the follow-up will follow the AASLD practice guideline for the management of hepatocellular carcinoma (2010)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhao, MD, Principal Investigator — Shandong Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] European Association for Study of Liver; European Organisation for Research and Treatment of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. Eur J Cancer. 2012 Mar;48(5):599-641. doi: 10.1016/j.ejca.2011.12.021. No abstract available. PMID 22424278
- [Background] Kobayashi M, Ikeda K, Hosaka T, Sezaki H, Someya T, Akuta N, Suzuki F, Suzuki Y, Saitoh S, Arase Y, Kumada H. Dysplastic nodules frequently develop into hepatocellular carcinoma in patients with chronic viral hepatitis and cirrhosis. Cancer. 2006 Feb 1;106(3):636-47. doi: 10.1002/cncr.21607. PMID 16369988
- [Background] Sato T, Kondo F, Ebara M, Sugiura N, Okabe S, Sunaga M, Yoshikawa M, Suzuki E, Ogasawara S, Shinozaki Y, Ooka Y, Chiba T, Kanai F, Kishimoto T, Nakatani Y, Fukusato T, Yokosuka O. Natural history of large regenerative nodules and dysplastic nodules in liver cirrhosis: 28-year follow-up study. Hepatol Int. 2015 Apr;9(2):330-6. doi: 10.1007/s12072-015-9620-6. Epub 2015 Mar 3. PMID 25788204
- [Background] Brenner H, Altenhofen L, Stock C, Hoffmeister M. Natural history of colorectal adenomas: birth cohort analysis among 3.6 million participants of screening colonoscopy. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1043-51. doi: 10.1158/1055-9965.EPI-13-0162. Epub 2013 Apr 30. PMID 23632815